CLINICAL TRIAL: NCT06998030
Title: Silent Threat: How Do Preoperative Albumin Levels Affect Outcomes in Geriatric Cancer Surgery
Brief Title: Silent Threat: Impact of Preoperative Albumin Levels on Outcomes in Geriatric Cancer Surgery
Status: Completed | Type: Observational
Sponsor: Dr Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Mustafa Kemal ŞAHİN, M.D, Dr Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital
Other Study IDs: 2025-03/53
Record Dates: First submitted 2025-05-13; First posted 2025-05-31 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Neoplasms; Aged; Hypoalbuminemia; Postoperative Complications; Malnutrition
MeSH Terms: conditions — Neoplasms; Hypoalbuminemia; Postoperative Complications; Malnutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1 (<3.5 g/dL, hypoalbuminemia): Participants with preoperative serum albumin levels less than 3.5 g/dL. This group represents geriatric cancer surgery patients who are considered to have hypoalbuminemia, indicating poor nutritional and/or inflammatory status prior to surgery.
- Group 2 (≥3.5 g/dL, normal): Participants with preoperative serum albumin levels equal to or greater than 3.5 g/dL. This group represents geriatric cancer surgery patients with normal preoperative albumin levels, reflecting adequate nutritional and inflammatory status prior to surgery.

SUMMARY:
This retrospective, single-center study aims to evaluate the impact of preoperative albumin levels on postoperative outcomes in geriatric patients (aged 65 and above) undergoing cancer surgery. The study will compare postoperative complication rates, length of hospital stay, and intensive care needs between patients with hypoalbuminemia and those with normal albumin levels.

DETAILED DESCRIPTION:
Malnutrition is a significant risk factor for postoperative complications in elderly cancer patients. Preoperative serum albumin is a key biomarker reflecting nutritional and inflammatory status. This study will retrospectively review the medical records of 330 geriatric patients (≥65 years) who underwent cancer surgery at Dr. Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital. Patients will be grouped according to preoperative albumin levels: Group 1 (<3.5 g/dL, hypoalbuminemia) and Group 2 (≥3.5 g/dL, normal). The primary aim is to compare postoperative complication rates, length of hospital stay, and intensive care requirements between these groups. The findings are expected to clarify the prognostic value of albumin and support individualized perioperative management in geriatric cancer surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 years or older
* Diagnosed with cancer and underwent cancer surgery
* Preoperative albumin level recorded before surgery

Exclusion Criteria:

* Preoperative sepsis, severe infection, or active inflammatory disease
* Emergency or palliative surgery
* Missing preoperative albumin value
* Incomplete medical records or follow-up data

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: This study will include geriatric patients aged 65 years and older who underwent elective cancer surgery at Dr. Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital. All participants must have a documented preoperative serum albumin level. Patients with emergency or palliative surgery, active infection or inflammatory disease, or missing/incomplete medical records will be excluded. The study population represents a real-world cohort of elderly cancer patients at increased risk for postoperative complications due to age-related physiological changes and comorbidities.
Sampling Method: Non-Probability Sample
Enrollment: 330 (Actual)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-05-10 (Actual)

PRIMARY OUTCOMES:
Postoperative Complication Rate | within 30 days after surgery
  The proportion of patients experiencing any postoperative complication (including but not limited to pulmonary complications, infections, or other adverse events) within 30 days after surgery, as assessed by clinical records and standardized criteria (e.g., Clavien-Dindo classification)

SECONDARY OUTCOMES:
Length of Hospital Stay | postoperative first 30 days
  Total number of days from the date of surgery to hospital discharge.
Postoperative Intensive Care Unit (ICU) Admission | immediately after the surgery
  The proportion of patients requiring ICU admission after surgery
Length of ICU Stay | 30 days after surgery
  The total duration of ICU stay following surgery
30-day Postoperative Mortality | within 30 days after surgery
  All-cause mortality within 30 days after surgery
Incidence of Specific Postoperative Pulmonary Complications | 30 days after surgery
  The number of patients developing pulmonary complications (e.g., pneumonia, pleural effusion, atelectasis, ARDS, respiratory failure) within 30 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa Kemal SAHIN, Principal Investigator — MUSTAFA KEMAL SAHİN
Locations (1):
- Dr. Abdurrahman Yurtaslan Ankara Oncology Education and Research Hospital Clinic of Anesthesiology and Reanimation, Ankara, Yenimahalle, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Song S, Qiu P, Wang H, Zhang D, Qi Q, Feng L. Low preoperative serum prealbumin levels and risk of postoperative complications after transsphenoidal surgery in nonfunctioning pituitary adenoma. Neurosurg Focus. 2022 Dec;53(6):E6. doi: 10.3171/2022.9.FOCUS22211. PMID 36455266
- [Background] Caras RJ, Lustik MB, Kern SQ, McMann LP, Sterbis JR. Preoperative Albumin Is Predictive of Early Postoperative Morbidity and Mortality in Common Urologic Oncologic Surgeries. Clin Genitourin Cancer. 2017 Apr;15(2):e255-e262. doi: 10.1016/j.clgc.2016.09.008. Epub 2016 Sep 23. PMID 27765612
- [Background] Loftus TJ, Brown MP, Slish JH, Rosenthal MD. Serum Levels of Prealbumin and Albumin for Preoperative Risk Stratification. Nutr Clin Pract. 2019 Jun;34(3):340-348. doi: 10.1002/ncp.10271. Epub 2019 Mar 25. PMID 30908744
- [Background] Heise D, Bednarsch J, Kroh A, Schipper S, Eickhoff R, Lang S, Neumann U, Ulmer F. Operative Time, Age, and Serum Albumin Predict Surgical Morbidity After Laparoscopic Liver Surgery. Surg Innov. 2021 Dec;28(6):714-722. doi: 10.1177/1553350621991223. Epub 2021 Feb 10. PMID 33568020